CLINICAL TRIAL: NCT02157792
Title: An Open-Label, First-in-Human Study of the Safety, Tolerability, and Pharmacokinetics of VX-970/M6620 in Combination With Cytotoxic Chemotherapy in Participants With Advanced Solid Tumors
Brief Title: M6620 First in Human Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS201923_0001; VX12-970-001 (Other: Other); 2012-003126-25 (EudraCT Number)
Record Dates: First submitted 2014-06-01; First posted 2014-06-06 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Advanced Solid Tumor
Keywords: Solid Tumor; Advanced Solid Tumor; VX12-970-001; M6620; VX-970; Gemcitabine; Cisplatin; Etoposide; Carboplatin; Irinotecan
MeSH Terms: interventions — berzosertib; Gemcitabine; Cisplatin; Etoposide; Carboplatin; Irinotecan

ARMS (6):
- Part A (Experimental): This part will be 3 + 3 dose escalation study of M6620 in combination with gemcitabine as well as gemcitabine and cisplatin in participants with advanced solid tumors.
  Interventions: Drug: M6620; Drug: Gemcitabine; Drug: Cisplatin
- Part B (Experimental): This part will be 3 + 3 dose escalation study of M6620 in combination with cisplatin or cisplatin and etoposide in participants with advanced solid tumors.
  Interventions: Drug: M6620; Drug: Cisplatin; Drug: Etoposide
- Part B2 (Experimental): This part will be 3 + 3 dose escalation study of M6620 in combination with irinotecan in participants with advanced solid tumors.
  Interventions: Drug: M6620; Drug: Irinotecan
- Part C1 (Experimental): This will be the expansion part of the study in which participants with advanced non-small cell lung cancer (NSCLC) will be administered M6620 in combination with gemcitabine.
  Interventions: Drug: M6620; Drug: Gemcitabine
- Part C2 (Experimental): This will be the expansion part of the study in which participants with advanced triple negative breast cancer (TNBC) will be administered M6620 in combination with cisplatin.
  Interventions: Drug: M6620; Drug: Cisplatin
- Part C3 (Experimental): This will be the expansion part of the study in which participants with platinum-resistant advanced small cell lung cancer (SCLC) will be administered M6620 in combination with cisplatin or carboplatin.
  Interventions: Drug: M6620; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: M6620
  Other Names: VX-970
Drug: Gemcitabine
  Arms: Part A; Part C1
Drug: Cisplatin
  Arms: Part A; Part B; Part C2; Part C3
Drug: Etoposide
  Arms: Part B
Drug: Carboplatin
  Arms: Part C3
Drug: Irinotecan
  Arms: Part B2

SUMMARY:
An Open-Label, First-in-Human Study of the Safety, Tolerability, and Pharmacokinetics (PK) of M6620 in Combination With Cytotoxic Chemotherapy in Participants With Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

Disease status

* Parts A and B/B2: Histologically or cytologically confirmed advanced solid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective, or for whom regimens containing gemcitabine, cisplatin, etoposide, and/or irinotecan might be considered, and with measurable disease according to RECIST criteria
* Part C1:

For Pre-screening:

* Advanced (metastatic or locally-advanced unresectable and not eligible for definitive treatment, e.g., surgery/radiotherapy), histologically confirmed non-small cell lung cancer (NSCLC)
* Available historical tumor specimen at the time of pre-screening or willing to provide a tumor biopsy (core) if the biopsy may be considered as part of standard clinical practice for the participant
* Received or did not tolerate standard approved targeted therapy, if appropriate for tumor genotype

For Screening:

* Measurable disease according to RECIST criteria

  -Part C2:
* Advanced (locally-advanced incurable or metastatic) histologically confirmed estrogen receptor, progesterone receptor, and human epidermal growth factor receptor 2 (HER2) negative breast cancer.
* Adequate available historical tumor specimen or willing to provide a tumor biopsy (core) if the biopsy may be considered as part of standard clinical practice for the participant
* Measurable disease according to RECIST criteria

  -Part C3:
* Advanced (locally-advanced incurable or metastatic) histologically confirmed SCLC that is platinum-resistant, defined as disease progression during initial treatment with a platinum-based regimen or progression within 90 days of completion of platinum therapy. Participants with platinum-resistant disease may receive a second-line non-platinum-based chemotherapy and subsequently be enrolled to this study. Participants who received and are resistant to a second-line platinum-based chemotherapy may also be enrolled into the study.
* Adequate available historical tumor specimen or willing to provide a tumor biopsy (core) if the biopsy may be considered as part of standard clinical practice for the participant
* Measurable disease according to RECIST criteria
* WHO performance status of 0 or 1
* Life expectancy of >=12 week
* Hematological and biochemical indices within protocol specified ranges at screening.

Exclusion Criteria:

* Radiotherapy (except for palliative reasons) endocrine therapy, immunotherapy, or chemotherapy during the previous 4 weeks (6 weeks for nitrosoureas and Mitomycin-C, and 4 weeks for investigational medicinal products) or less than 4 drug half-lives, whichever greater, before first dose of study drug.
* Parts A, B and B2:

  * Greater than 6 cycles of prior treatment with cisplatin and/or carboplatin.

    1. Part A/B: History of prior dose reductions or dose interruptions while receiving cisplatin or carboplatin due to toxicity from the platinum or intolerance to either agent.
    2. Part B2: Prior exposure to irinotecan is permitted except for participants with a known hypersensitivity reaction to irinotecan.
  * Participants with a known history of Grade 4 thrombocytopenia or Grade 4 neutropenia while receiving prior therapy.
* Part C1:

  * Any cytotoxic chemotherapy beyond 1 line of platinum-based chemotherapy. One additional line of non-platinum based therapy in the advanced setting

    1. Pre-screening Only*: Participants may currently be receiving platinum-based chemotherapy in the advanced setting, or have completed 1 line of platinum-based chemotherapy and are currently receiving a second-line non-platinum-based therapy or maintenance therapy
    2. There is no restriction on prior immunotherapy or targeted therapy unless combined together with a cytotoxic agent
  * Any prior gemcitabine for the treatment of NSCLC in any setting within 6 months
  * Participants who are known to be TP53 wild-type, unless they are determined to have ATM loss of expression during screening or pre-screening or until all the planned participants with TP53 mutation are enrolled as determined by the medical monitor
  * Participants with unknown TP53 mutational status will be enrolled until the group of approximately 10 participants without TP53 mutation or until all the planned participants with TP53 mutation are enrolled as determined by the medical monitor
* Part C2:

  * Any prior platinum therapy in the adjuvant or neoadjuvant within 6 months of screening
  * Relapse within 3 months of completion of prior adjuvant or neoadjuvant chemotherapy
  * Any prior chemotherapy in the metastatic setting with the exception of either a taxane or an anthracycline in the first-line metastatic setting

    (a) There is no restriction on prior immunotherapy or targeted therapy in the metastatic setting unless combined together with a cytotoxic agent
  * Participants with known BRCA1/BRCA2 germline mutations, either determined and documented prior to Screening, or determined during Screening. Participants with unknown BRCA1/BRCA2 status may be enrolled at discretion of the sponsor
  * Participants who are documented to be non-basaloid subtype using molecular profiling assay (e.g. PAM50 assay) prior to Screening
  * Participants with unknown BRCA1/BRCA2 or basaloid subtype status will be enrolled until the number of enrolled participant is approximately 40. If approximately 40 participants have been enrolled and a minimum of 30 participants who are basaloid positive and BRCA1/BRCA2 germline wild-type have not been enrolled, the basaloid subtype and BRCA status assay will be required at Screening to exclude participants who are basaloid negative or have BRCA1/BRCA2 germline mutations.
* Part C3:

  * Prior platinum-sensitive participants , unless they progress on or within 90 days of completion of platinum-based regimen
  * There is no restriction on prior immunotherapy or targeted therapy in the metastatic setting unless combined together with a cytotoxic agent
  * During prior carboplatin therapy, requirement for dose reduction below AUC 5 mg.min/mL or discontinuation of carboplatin for toxicity or lack of tolerability.
* Unresolved toxicity of Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or greater from previous anti-cancer therapy or radiotherapy
* History of spinal cord compression or brain metastases, unless asymptomatic, treated, stable, and not requiring treatment with steroids for at least 4 weeks before first dose of study drug. Any history of leptomeningeal metastases.
* Female participants who are already pregnant or lactating, or plan to become pregnant within 6 months of the last dose of study drug are excluded. Female participants of childbearing potential must adhere to contraception guidelines
* Male participants with partners of child-bearing potential must agree to adhere to contraception guidelines. Men with pregnant or lactating partners or partners who plan to become pregnant during the study or within 6 months of the last dose of study drug are excluded
* Serious cardiac or other co-morbid disease, as specified in the protocol
* Prior bone marrow transplant or extensive radiotherapy to greater than 15% of bone marrow
* Part C:

  * Current malignancies of other types, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin
* Major surgery =<2 weeks before starting study drug, or incomplete recovery from a prior major surgical procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-12-10 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Parts A, B, B2, C1, C2, C3: Safety parameters, including adverse event (AEs), clinical laboratory values (serum chemistry, hematology, and urinalysis), vital signs, and electrocardiogram (ECG) assessments | Screening through Safety Follow-up (approximately 22 weeks)
Parts C1, C2, C3: Overall Response Rate (ORR) for all participants in Part C1 (NSCLC), ORR for participants in Part C2 (TNBC) who are basaloid subtype and BRCA1/BRCA2 germline wild-type, ORR for all participants in Part C3 (SCLC) | 1 year

SECONDARY OUTCOMES:
Part A: Maximum tolerated dose (MTD) of M6620 administered in combination with cisplatin and gemcitabine and in combination with gemcitabine | 1 year
Part A: Pharmacokinetic (PK) parameter estimates of M6620 in combination with cisplatin and gemcitabine and in combination with gemcitabine | 1 year
Part B, B2: Maximum tolerated dose (MTD) of M6620 in combination with cisplatin or cisplatin and etoposide or irinotecan | 1 year
Part B, B2: PK parameter estimates of M6620 in combination with cisplatin or cisplatin and etoposide or irinotecan | 1 year
Part B: PK parameter estimates of etoposide derived from plasma concentration-time data after coadministration with M6620 and in the absence of M6620 | 1 year
Parts A, B, B2: Objective tumor response (OR) as evaluated by Response Criteria Evaluation in Solid Tumors (RECIST) 1.1 | 1 year
Part C2: Overall Response Rate in all participants in Part C2 | 1 year
Parts C1, C2, C3: Progression Free Survival (PFS) | 1 year
Parts C1, C2, C3: Response Duration (RD) | 1 year
Parts C1, C2, C3: Overall Survival (OS) | 1 year
Parts C1, C2, C3: Clinical benefit (Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) of 6 months or greater) | 1 year
Parts C1, C2, C3: PK parameter estimates of M6620 including maximum concentrations (Cmax), area under the curve (AUC), apparent volume at steady state (Vss), clearance (CL) and terminal elimination half-life (t1/2) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc., a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (31):
- United States (24):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Sharp Memorial Hospital, San Diego, California
  - Stanford, California
  - Rocky Mountain Cancer Centers, LLP, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Northwestern Center for Clinical Research, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Breslin Cancer Center, Lansing, Michigan
  - University Of Minnesota Hospital, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Hackensack University Medical Center PARTNER, Hackensack, New Jersey
  - Long Island Jewish Medical Center - Monter Cancer Center, Lake Success, New York
  - University Hospitals Case Medical Center - Case Comprehensive Cancer Center at, Cleveland, Ohio
  - OSU - James Comprehensive Cancer Center - Division of Hematology, Columbus, Ohio
  - Greenville Health System, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - US Oncology - Texas Oncology-Midtown - Austin Midtown, Austin, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - University of Texas M. D. Anderson Cancer Center - Investigational Cancer Therapeutics - Partner, Houston, Texas
  - Texas Oncology San Antonio Medical Cente, San Antonio, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates - Hampton, Norfolk, Virginia
  - Northwest Cancer Specialists , P.C., Vancouver, Washington
- United Kingdom (7):
  - Freeman Hospital - PARENT, Newcastle upon Tyne, England
  - Churchill Hospital - PARENT, Oxford, England
  - Beatson West of Scotland Cancer Centre - Dept of Medical Oncology, Glasgow, Scotland
  - Royal Marsden Hospital - Dept of Oncology, Sutton, Surrey
  - Guy's Hospital - PARENT, London
  - Sarah Cannon Research Institute UK, London
  - The Christie - Dept of Oncology, Manchester

REFERENCES:
- [Derived] Middleton MR, Dean E, Evans TRJ, Shapiro GI, Pollard J, Hendriks BS, Falk M, Diaz-Padilla I, Plummer R. Phase 1 study of the ATR inhibitor berzosertib (formerly M6620, VX-970) combined with gemcitabine +/- cisplatin in patients with advanced solid tumours. Br J Cancer. 2021 Aug;125(4):510-519. doi: 10.1038/s41416-021-01405-x. Epub 2021 May 26. PMID 34040175
- [Derived] Shapiro GI, Wesolowski R, Devoe C, Lord S, Pollard J, Hendriks BS, Falk M, Diaz-Padilla I, Plummer R, Yap TA. Phase 1 study of the ATR inhibitor berzosertib in combination with cisplatin in patients with advanced solid tumours. Br J Cancer. 2021 Aug;125(4):520-527. doi: 10.1038/s41416-021-01406-w. Epub 2021 May 26. PMID 34040174
- [Derived] Terranova N, Jansen M, Falk M, Hendriks BS. Population pharmacokinetics of ATR inhibitor berzosertib in phase I studies for different cancer types. Cancer Chemother Pharmacol. 2021 Feb;87(2):185-196. doi: 10.1007/s00280-020-04184-z. Epub 2020 Nov 4. PMID 33145616